CLINICAL TRIAL: NCT04757961
Title: Evaluation of an ACT-based Narrative Intervention for Individuals Taking Antidepressant Medication
Brief Title: Evaluation of an Acceptance and Commitment Therapy-Based Narrative Intervention for Individuals Taking Antidepressants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Responsible Party: Principal Investigator, Michael Levin, Associate Professor, Utah State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 11523
Record Dates: First submitted 2021-02-11; First posted 2021-02-17 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Depressive Symptoms
Keywords: ACT; narrative intervention; story-telling intervention; depression; antidepressant
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned with equal likelihood to receive the online ACT-based intervention (LifeStories) or the waitlist control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestories (Experimental): Participants in this condition will be actively participating in the online intervention for 4 weeks.
  Interventions: Behavioral: LifeStories
- Waitlist Control Condition (No Intervention): Participant in the waitlist group will be asked to not use other self-help websites or books for four weeks, after which they will be given weekly access to LifeStories modules. All participants will be asked to continue their antidepressant treatment as usual as directed by their primary care provider.

INTERVENTIONS:
Behavioral: LifeStories — The content of LifeStories is divided thematically into core ACT concepts across the four episodes as follows: 1) cultivating awareness of the transient nature of mood experiences and the benefit of trying out various strategies to cope with depression when it arises; 2) clarifying one's own values and setting personal goals related to these values; 3) developing a more accepting and nonjudgmental stance towards difficult thoughts and feelings and practicing self-compassion;and 4) living more mindfully in the present moment.
  Arms: Lifestories

SUMMARY:
This study aims to compare the efficacy of LifeStories on depression symptomatology compared to antidepressant treatment alone, in addition to examining the effect of the intervention on health-related quality of life. Participants will be randomly assigned to either an online ACT-based narrative intervention (Lifestories) or the waitlist control condition (antidepressant treatment alone). It is hypothesized that participants who receive the LifeStories will result in decreased depression and increased quality of life, general functioning and decreased psychological inflexibility compared to the waitlist group.

DETAILED DESCRIPTION:
The purpose of this study is to test the efficacy of an online, self-guided ACT-based narrative intervention for adults currently taking antidepressant medication. To test the effects of LifeStories on depression severity, quality of life, general functioning and psychological inflexibility, the investigators will conduct a randomized controlled trial with two conditions (LifeStories and waitlist control) using a sample of 90 adults currently taking antidepressant medication. Interested individuals will complete a screening survey to determine eligibility. After being informed about the study and potential risks, eligible participants who provide informed consent will be asked to complete a baseline survey. Participants will then be randomized to LifeStories or a waitlist control conditions, each lasting 4 weeks. Those in the waitlist group will be asked to not use other self-help websites or books for four weeks, after which they will be given weekly access to LifeStories modules. Participants in both groups will be asked to complete a midtreatment survey 2 weeks after baseline, and a posttreatment survey 4 weeks after baseline (i.e. after completing the 4-week video intervention for those in the active condition).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Currently residing in the United States
3. Currently taking antidepressant medication prescribed by a primary care provider (PCP)
4. Meets criteria for at least moderate depression on the 9-item Patient Health Questionnaire
5. Fluent in English
6. Reliable access to an internet browser, and internet speed that is sufficient for streaming online videos

Exclusion Criteria:

1. Change in medication regimen in past 6 weeks
2. Presently seeing a mental health specialist (e.g. psychologist, psychiatrist, counselor, social worker)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Change in depression severity | Baseline, Mid-treatment (2 weeks post baseline), Post-treatment (4 weeks post baseline)
  Patient Health Questionnaire 9-item (PHQ-9; Kroenke et al., 2001): The PHQ is a 9-item measure of depression severity, which asks respondents to report their frequency of depressive symptoms over the past two weeks, rated from 0 "not at all" to 3 "nearly every day". The PHQ-9 provides a total score which indicates current depression severity according to the following levels: minimal, mild, moderate, moderately severe, and severe. Higher scores indicate higher depression.

SECONDARY OUTCOMES:
Change in health-related quality of life | Baseline, Mid-treatment (2 weeks post baseline), Post-treatment (4 weeks post baseline)
  Short Form Health Survey (SF-12; Ware et al., 1996): The SF-12 is a 12-item measure of quality of life and general functioning. Respondents are asked to rate their present level of health or emotion-related impairment in daily activities. Items are rated on a scale from 1 "all of the time" to 6 "none of the time," with higher scores indicating greater health-related quality of life.
Change in psychological inflexibility | Baseline, Mid-treatment (2 weeks post baseline), Post-treatment (4 weeks post baseline)
  Acceptance and Action Questionnaire-II (AAQ-II; Bond et al., 2011): The AAQ-II is a 10-item measure of psychological inflexibility and experiential avoidance. Items are rated on a 7-point scale ranging from 1 "never true" to 7 "always true." A total score is calculated by reverse coding so that higher scores indicate greater psychological flexibility.

OTHER OUTCOMES:
Changes in treatment preferences | Baseline, Post-treatment (4 weeks post baseline)
  General Help Seeking Questionnaire (GHSQ; Wilson, Deane, Ciarocchi, & Rickwood): We will use an adapted version of the GHSQ which is a validated measure of help-seeking intentions from a variety of formal (e.g. psychologist, PCP) and informal (e.g. friends, family) supports, rated on a 7-point scale from 1 "extremely likely" to 7 "extremely unlikely," with higher scores on each item indicating greater likelihood of seeking help from that source.
Treatment adherence | Post-treatment (4 weeks post baseline)
  Participants will be asked to rate their adherence to the homework exercises from the online program on a 7-point scale from 1 "did no recommended assignments" to 7 "did all recommended assignments," using a scale adapted from previous self-help studies (Abramowitz, Moore, Braddock, & Harrington, 2009). Higher scores on this measure indicate greater treatment adherence.
Treatment satisfaction | Post-treatment (4 weeks post baseline)
  System Usability Scale (SUS; Brooke, 1996): The SUS is a 10-item measure of usability and satisfaction with programs with established reliability and validity (Lewis, 2009). Items on the SUS are rated on a scale from 1 "strongly disagree" to 5 "strongly disagree, with higher scores indicating greater treatment satisfaction. We will additionally ask those in the active condition a series of free-response questions assessing their favorite and least favorite aspects of LifeStories, as well as their perspectives on how using the program may have helped them manage depression.
Changes in treatment utilization | Baseline, post-treatment (4 weeks post baseline)
  We will ask participants at baseline and post-treatment a series of yes/no questions that we constructed which ask if they are engaged in treatment with a mental health specialist, are planning to see a mental health specialist, or have made any recent changes to their antidepressant treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Levin, Ph.D, Principal Investigator — Utah State University
Locations (1):
- Utah State University, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abramowitz JS, Moore EL, Braddock AE, Harrington DL. Self-help cognitive-behavioral therapy with minimal therapist contact for social phobia: a controlled trial. J Behav Ther Exp Psychiatry. 2009 Mar;40(1):98-105. doi: 10.1016/j.jbtep.2008.04.004. Epub 2008 Apr 26. PMID 18514614
- [Background] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Wilson, C.J., Deane, F.P., Ciarrochi, J. & Rickwood, D. (2005). Measuring help-seeking intentions: Properties of the General Help-Seeking Questionnaire. Canadian Journal of Counselling, 39(1), 15-28.
- [Background] Brooke, J. (1996). SUS: A "Quick and Dirty" Usability Scale. In: Jordan, P.W., Thomas, B., Weerdmeester, B.A., McClelland (eds.) Usability Evaluation in Industry, pp. 189-194. Taylor & Francis, London.
- [Background] Levin, M. E., Stocke, K., Pierce, B., & Levin, C. (2018). Do college students use online self-help? A survey of intentions and use of mental health resources. Journal of college student psychotherapy, 32(3), 181-198.
- [Background] Lewis, J. R., & Sauro, J. (2009, July). The factor structure of the system usability scale. In International Conference on Human Centered Design (pp. 94-103). Springer, Berlin, Heidelberg.
- [Derived] Davis CH, Donahue ML, Gaudiano BA, Uebelacker LA, Twohig MP, Levin ME. Adding online storytelling-based acceptance and commitment therapy to antidepressant treatment for primary care patients: a randomized clinical trial. Cogn Behav Ther. 2024 Jan;53(1):48-69. doi: 10.1080/16506073.2023.2265560. Epub 2024 Jan 2. PMID 37855277